CLINICAL TRIAL: NCT02271984
Title: A Phase I, Open-Label, Randomized, Single Dose, Five Period, Crossover, Single Center Trial To Assess The Relative Bioavailability Of The 150 mg ODT Formulation Of L PZQ (MSC2499550A) Versus The Current 500 mg PZQ Commercial Racemate Tablet Formulation In Healthy Male Volunteers
Brief Title: Relative Bioavailability Trial of L-Praziquantel in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 200661-001
Record Dates: First submitted 2014-10-20; First posted 2014-10-22 (Estimated); Results first posted 2018-01-03 (Actual); Last update posted 2018-01-03 (Actual); Status verified 2017-05

CONDITIONS: Healthy
Keywords: Healthy; Praziquantel; L-PZQ; PZQ; MSC2499550A; Bioavailability; Pharmacokinetics
MeSH Terms: interventions — Praziquantel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- Treatment A: MSC2499550A (Experimental): MSC2499550A: 20 milligram per kilogram (mg/kg) under fed condition
  Interventions: Drug: MSC2499550A
- Treatment B: Cysticide (Experimental): Cysticide® 40 mg/kg under fed condition
  Interventions: Drug: Cysticide
- Treatment C: MSC2499550A (Experimental): C1:MSC2499550A :10 mg/kg under fed condition C2:MSC2499550A : 30 mg/kg under fed condition
  Interventions: Drug: MSC2499550A
- Treatment D: MSC2499550A (Experimental): MSC2499550A 20 mg/kg under fasting condition
  Interventions: Drug: MSC2499550A
- Treatment E: MSC2499550A (Experimental): MSC2499550A: 20 mg/kg directly disintegrated in mouth under fed condition
  Interventions: Drug: MSC2499550A

INTERVENTIONS:
Drug: MSC2499550A — Subjects will receive a single oral dose of MSC2499550A formulation at 20 mg/kg dispersed in water under fed condition in one of the intervention periods. There will be a wash-out period of at least 7 days between each intervention period.
  Other Names: L-PZQ
  Arms: Treatment A: MSC2499550A
Drug: Cysticide — Subjects will receive a single oral dose of current PZQ formulation (Cysticide®) at 40 mg/kg with water, under fed condition in one of the intervention periods. There will be a wash-out period of at least 7 days between each of the intervention period.
  Other Names: Praziquantel
  Arms: Treatment B: Cysticide
Drug: MSC2499550A — Subjects will receive a single oral dose of MSC2499550A formulation at 10 mg/kg dispersed in water under fed condition in one of the intervention periods. There will be a wash-out period of at least 7 days between each of the intervention period.
  Other Names: L-PZQ
  Arms: Treatment C: MSC2499550A
Drug: MSC2499550A — Subjects will receive a single oral dose of MSC2499550A formulation at 30 mg/kg dispersed in water under fed condition in one of the intervention periods. There will be a wash-out period of at least 7 days between each of the intervention period.
  Other Names: L-PZQ
  Arms: Treatment C: MSC2499550A
Drug: MSC2499550A — Subjects will receive a single oral dose of MSC2499550A formulation at 20 mg/kg dispersed in water in fasted condition in one of the intervention periods. There will be a wash-out period of at least 7 days between each of the intervention period.
  Other Names: L-PZQ
  Arms: Treatment D: MSC2499550A
Drug: MSC2499550A — Subjects will receive a single oral dose of MSC2499550A formulation at 20 mg/kg directly disintegrated in the mouth without water under fed conditions in one of the intervention periods. There will be a wash-out period of at least 7 days between each of the intervention period.
  Other Names: L-PZQ
  Arms: Treatment E: MSC2499550A

SUMMARY:
This is a phase I, open-label, randomized, 5 period, crossover, single-center trial. The purpose of this trial is to assess the relative bio-availability of L-praziquantel (L-PZQ [MSC2499550A]) oral dispersible tablet (ODT) formulation (150 milligram [mg]) versus the current marketed racemate praziquantel (PZQ) (Cysticide® 500 mg) formulation in healthy male volunteers under fed conditions.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males aged 18-55 years of age (inclusive at screening)
* Male subjects with partners of childbearing potential must have had a vasectomy or use acceptable methods of birth control (that is, condoms) and not donate sperm during, and until 90 days after the last dose of the trial medication
* Written informed consent prior to any trial related procedure
* Have a body weight of greater than or equal to (>=) 55.0 kilogram (kg) to less than (<) 95.0 kg and a body mass index (BMI) of 18.5 to 29.9 kilogram per square meter (kg/m^2) (inclusive)
* Able to communicate well with the Investigator, understanding the protocol requirements and restrictions, and willing to comply with the requirements of the entire trial
* Non-smoker (= 0 cigarettes, pipes, cigars or others) since at least 3 months
* Electrocardiogram (ECG) recording (12-lead) without signs of clinically relevant pathology in particular corrected QT Interval (QTc) (Bazett) < 450 milliseconds (ms)
* Vital signs (systolic and diastolic blood pressure, pulse) in supine position and body temperature within the normal range or showing no clinically relevant deviation as judged by the medical Investigator

Exclusion Criteria:

* Any surgical or medical condition, including findings in the medical history or in the prestudy assessments, or any other significant disease, that in the opinion of the Investigator, constitutes a risk or a contraindication for the participation of the subject in the study or that could interfere with the study objectives, conduct or evaluation
* History of surgery of the gastrointestinal tract (GI), history of other GI tract diseases, or acute GI tract infections in the last 2 weeks, which could influence the GI absorption and/or motility according to the Investigator's opinion
* Any clinically relevant abnormality in the safety laboratory parameters as judged by the Investigator
* Have positive results from serology examination for Hepatitis B surface antigen (HBsAg), Hepatitis C Virus (HCV) or Human Immunodeficiency Virus (HIV)
* Allergy: ascertained or presumptive hypersensitivity to the active drug substance and/or formulations ingredients; history of anaphylaxis to drugs or allergic reactions in general, which the Investigator considers may affect the outcome of the trial
* History or presence of drug abuse (amphetamines, barbiturates, benzodiazepines, cocaine, opiates, phencyclidine (phenylcyclohexalpiperidine), tetrahydrocannabinol, tricyclic antidepressants, methadone, methamphetamine, oxycodone and propoxyphene) or alcohol abuse at screening and on each admission as defined by the Investigator
* Loss or donation of more than 400 milliliter (mL) of blood within 90 days prior to first praziquantel (PZQ) administration
* Administration of any investigational product or use of any investigational device within 60 days prior to first PZQ administration
* Subjects who have used drugs that may affect the pharmacokinetics (PK) of PZQ from 14 days before dosing until the last PK sample, for example, phenytoin, barbiturates, primidone, carbamazapine, oxcarbazepine, topiramate, felbamate, rifampicin, nelfinavir, ritonavir, griseofulvin, oral ketoconazole, on discretion of the Investigator
* Consumption of substances known to be potent inhibitors or inducers of cytochrome -P450 enzymes (CYP P450s) such as grapefruit juice, grapefruit juice containing products, and herbal remedies or dietary supplements containing St. John's Wort, in the 2 weeks before dosing
* Unlikely to comply with the protocol requirements, instructions and trial-related restrictions, for example, uncooperative attitude, inability to return for follow-up visits, and improbability of completing the trial
* Non-acceptance of study breakfast (for example, vegetarians, vegans and subjects who follow special diets)
* Excessive consumption of beverages -containing xanthine (> 5 cups ) of coffee a day, or equivalent or inability to stop consuming caffeine from 48 hours prior to drug administration until discharge from the clinic
* Subject is the Investigator or any Sub-Investigator, research assistant, pharmacist, trial coordinator, other staff or relative thereof directly involved in the conduct of the trial
* Vulnerable subjects (for example, persons kept in detention)
* Legal incapacity or limited legal capacity

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2014-10-31 (Actual); Primary Completion 2014-12-31 (Actual); Study Completion 2014-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Responsible, Study Director — Merck KGaA, Darmstadt, Germany
Locations (1):
- Please contact the Merck KGaA Communication Center, Darmstadt, Germany

REFERENCES:
- [Derived] Bagchus WM, Bezuidenhout D, Harrison-Moench E, Kourany-Lefoll E, Wolna P, Yalkinoglu O. Relative Bioavailability of Orally Dispersible Tablet Formulations of Levo- and Racemic Praziquantel: Two Phase I Studies. Clin Transl Sci. 2019 Jan;12(1):66-76. doi: 10.1111/cts.12601. Epub 2018 Dec 21. PMID 30536632

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Subjects were randomized to receive a sequence of 5 treatments over 5 treatment periods. A total of 36 were enrolled subjects, three in each of the 12 possible sequences were distributed.
Groups:
- ABC1DE: Subjects received a single oral dose of MSC2499550A oral disintegrating tablet (ODT) formulation at 20 milligram per kilogram (mg/kg) dispersed in water (A) in first intervention period followed by single oral dose of current PZQ formulation (Cysticide®) at 40 mg/kg with water (B) in second intervention period followed by a single oral dose of MSC2499550A formulation at 10 mg/kg dispersed in water (C1) in third intervention period under fed conditions followed by a single oral dose of MSC2499550A formulation at 20 mg/kg dispersed in water (D) in fourth intervention period under fasted conditions followed by a single oral dose of MSC2499550A formulation at 20 mg/kg directly disintegrated in the mouth (E) in fifth intervention period under fed condition. There was a wash-out period of at least 7 days between each intervention period.
- ABDEC1: Subjects received a single oral dose of MSC2499550A ODT formulation at 20 mg/kg dispersed in water (A) in first intervention period followed by single oral dose of current PZQ formulation (Cysticide®) at 40 mg/kg with water (B) in second intervention period under fed condition followed by a single oral dose of MSC2499550A formulation at 20 mg/kg dispersed in water (D) in third intervention period under fasted conditions followed by a single oral dose of MSC2499550A formulation at 20 mg/kg directly disintegrated in the mouth (E) in fourth intervention period followed by a single oral dose of MSC2499550A formulation at 10 mg/kg dispersed in water (C1) in fifth intervention period under fed conditions. There was a wash-out period of at least 7 days between each intervention period.
- ABEC1D: Subjects received a single oral dose of MSC2499550A ODT formulation at 20 mg/kg dispersed in water (A) in first intervention period followed by single oral dose of current PZQ formulation (Cysticide®) at 40 mg/kg with water (B) in second intervention period followed by a single oral dose of MSC2499550A formulation at 20 mg/kg directly disintegrated in the mouth (E) in third intervention period followed by a single oral dose of MSC2499550A formulation at 10 mg/kg dispersed in water (C1) in fourth intervention period under fed conditions followed by a single oral dose of MSC2499550A formulation at 20 mg/kg dispersed in water (D) in fifth intervention period under fasted conditions. There was a wash-out period of at least 7 days between each intervention period.
- BAC1DE: Subjects received a single oral dose of current PZQ formulation (Cysticide®) at 40 mg/kg with water (B) in first intervention period followed by a single oral dose of MSC2499550A ODT formulation at 20 mg/kg dispersed in water (A) in second intervention period followed by a single oral dose of MSC2499550A formulation at 10 mg/kg dispersed in water (C1) in third intervention period under fed conditions followed by a single oral dose of MSC2499550A formulation at 20 mg/kg dispersed in water (D) in fourth intervention period under fasted conditions followed by a single oral dose of MSC2499550A formulation at 20 mg/kg directly disintegrated in the mouth (E) in fifth intervention period under fed condition. There was a wash-out period of at least 7 days between each intervention period.
- BADEC1: Subjects received a single oral dose of current PZQ formulation (Cysticide®) at 40 mg/kg with water (B) in first intervention period followed by a single oral dose of MSC2499550A ODT formulation at 20 mg/kg dispersed in water (A) in second intervention period under fed conditions followed by a single oral dose of MSC2499550A formulation at 20 mg/kg dispersed in water (D) in third intervention period under fasted conditions followed by a single oral dose of MSC2499550A formulation at 20 mg/kg directly disintegrated in the mouth (E) in fourth intervention period followed by a single oral dose of MSC2499550A formulation at 10 mg/kg dispersed in water (C1) in fifth intervention period under fed conditions. There was a wash-out period of at least 7 days between each intervention period.
- BAEC1D: Subjects received a single oral dose of current PZQ formulation (Cysticide®) at 40 mg/kg with water (B) in first intervention period followed by a single oral dose of MSC2499550A ODT formulation at 20 mg/kg dispersed in water (A) in second intervention period followed by a single oral dose of MSC2499550A formulation at 20 mg/kg directly disintegrated in the mouth (E) in third intervention period followed by a single oral dose of MSC2499550A formulation at 10 mg/kg dispersed in water (C1) in fourth intervention period under fed conditions followed by a single oral dose of MSC2499550A formulation at 20 mg/kg dispersed in water (D) in fifth intervention period under fasted conditions. There was a wash-out period of at least 7 days between each intervention period.
- ABC2DE: Subjects received a single oral dose of MSC2499550A ODT formulation at 20 mg/kg dispersed in water (A) in first intervention period followed by single oral dose of current PZQ formulation (Cysticide®) at 40 mg/kg with water (B) in second intervention period followed by a single oral dose of MSC2499550A formulation at 30 mg/kg dispersed in water (C2) in third intervention period under fed conditions followed by a single oral dose of MSC2499550A formulation at 20 mg/kg dispersed in water (D) in fourth intervention period under fasted conditions followed by a single oral dose of MSC2499550A formulation at 20 mg/kg directly disintegrated in the mouth (E) in fifth intervention period under fed condition. There was a wash-out period of at least 7 days between each intervention period.
- ABDEC2: Subjects received a single oral dose of MSC2499550A ODT formulation at 20 mg/kg dispersed in water (A) in first intervention period followed by single oral dose of current PZQ formulation (Cysticide®) at 40 mg/kg with water (B) in second intervention period under fed conditions followed by a single oral dose of MSC2499550A formulation at 20 mg/kg dispersed in water (D) in third intervention period under fasted conditions followed by a single oral dose of MSC2499550A formulation at 20 mg/kg directly disintegrated in the mouth (E) in fourth intervention period followed by a single oral dose of MSC2499550A formulation at 30 mg/kg dispersed in water (C2) in fifth intervention period under fed conditions. There was a wash-out period of at least 7 days between each intervention period.
- ABEC2D: Subjects received a single oral dose of MSC2499550A ODT formulation at 20 mg/kg dispersed in water (A) in first intervention period followed by single oral dose of current PZQ formulation (Cysticide®) at 40 mg/kg with water (B) in second intervention period followed by a single oral dose of MSC2499550A formulation at 20 mg/kg directly disintegrated in the mouth (E) in third intervention period followed by a single oral dose of MSC2499550A formulation at 30 mg/kg dispersed in water (C2) in fourth intervention period under fed conditions followed by a single oral dose of MSC2499550A formulation at 20 mg/kg dispersed in water (D) in fifth intervention period under fasted conditions. There was a wash-out period of at least 7 days between each intervention period.
- BAC2DE: Subjects received a single oral dose of current PZQ formulation (Cysticide®) at 40 mg/kg with water (B) in first intervention period followed by a single oral dose of MSC2499550A ODT formulation at 20 mg/kg dispersed in water (A) in second intervention period followed by a single oral dose of MSC2499550A formulation at 30 mg/kg dispersed in water (C2) in third intervention period under fed conditions followed by a single oral dose of MSC2499550A formulation at 20 mg/kg dispersed in water (D) in fourth intervention period under fasted conditions followed by a single oral dose of MSC2499550A formulation at 20 mg/kg directly disintegrated in the mouth (E) in fifth intervention period under fed condition. There was a wash-out period of at least 7 days between each intervention period.
- BADEC2: Subjects received a single oral dose of current PZQ formulation (Cysticide®) at 40 mg/kg with water (B) in first intervention period followed by a single oral dose of MSC2499550A ODT formulation at 20 mg/kg dispersed in water (A) in second intervention period under fed conditions followed by a single oral dose of MSC2499550A formulation at 20 mg/kg dispersed in water (D) in third intervention period under fasted conditions followed by a single oral dose of MSC2499550A formulation at 20 mg/kg directly disintegrated in the mouth (E) in fourth intervention period followed by a single oral dose of MSC2499550A formulation at 30 mg/kg dispersed in water (C2) in fifth intervention period under fed conditions. There was a wash-out period of at least 7 days between each intervention period.
- BAEC2D: Subjects received a single oral dose of current PZQ formulation (Cysticide®) at 40 mg/kg with water (B) in first intervention period followed by a single oral dose of MSC2499550A ODT formulation at 20 mg/kg dispersed in water (A) in second intervention period followed by a single oral dose of MSC2499550A formulation at 20 mg/kg directly disintegrated in the mouth (E) in third intervention followed by a single oral dose of MSC2499550A formulation at 30 mg/kg dispersed in water (C2) in fourth intervention under fed conditions followed by a single oral dose of MSC2499550A formulation at 20 mg/kg dispersed in water (D) in fifth intervention period under fasted conditions. There was a wash-out period of at least 7 days between each intervention period.
Period: First Intervention Period (1 Day)
Arm/Group | ABC1DE | ABDEC1 | ABEC1D | BAC1DE | BADEC1 | BAEC1D | ABC2DE | ABDEC2 | ABEC2D | BAC2DE | BADEC2 | BAEC2D
Started | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3
Completed | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Washout Period 1 (7 Days)
Arm/Group | ABC1DE | ABDEC1 | ABEC1D | BAC1DE | BADEC1 | BAEC1D | ABC2DE | ABDEC2 | ABEC2D | BAC2DE | BADEC2 | BAEC2D
Started | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3
Completed | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Second Intervention Period (1 Day)
Arm/Group | ABC1DE | ABDEC1 | ABEC1D | BAC1DE | BADEC1 | BAEC1D | ABC2DE | ABDEC2 | ABEC2D | BAC2DE | BADEC2 | BAEC2D
Started | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3
Completed | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Washout Period 2 (7 Days)
Arm/Group | ABC1DE | ABDEC1 | ABEC1D | BAC1DE | BADEC1 | BAEC1D | ABC2DE | ABDEC2 | ABEC2D | BAC2DE | BADEC2 | BAEC2D
Started | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3
Completed | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Third Intervention Period (1 Day)
Arm/Group | ABC1DE | ABDEC1 | ABEC1D | BAC1DE | BADEC1 | BAEC1D | ABC2DE | ABDEC2 | ABEC2D | BAC2DE | BADEC2 | BAEC2D
Started | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3
Completed | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Washout Period 3 (7 Days)
Arm/Group | ABC1DE | ABDEC1 | ABEC1D | BAC1DE | BADEC1 | BAEC1D | ABC2DE | ABDEC2 | ABEC2D | BAC2DE | BADEC2 | BAEC2D
Started | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3
Completed | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Fourth Intervention Period (Day 1)
Arm/Group | ABC1DE | ABDEC1 | ABEC1D | BAC1DE | BADEC1 | BAEC1D | ABC2DE | ABDEC2 | ABEC2D | BAC2DE | BADEC2 | BAEC2D
Started | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3
Completed | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Washout Period 4 (7 Days)
Arm/Group | ABC1DE | ABDEC1 | ABEC1D | BAC1DE | BADEC1 | BAEC1D | ABC2DE | ABDEC2 | ABEC2D | BAC2DE | BADEC2 | BAEC2D
Started | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3
Completed | 3 | 3 | 3 | 3 | 3 | 2 | 3 | 2 | 3 | 3 | 3 | 3
Not Completed | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Period: Fifth Intervention Period (1 Day)
Arm/Group | ABC1DE | ABDEC1 | ABEC1D | BAC1DE | BADEC1 | BAEC1D | ABC2DE | ABDEC2 | ABEC2D | BAC2DE | BADEC2 | BAEC2D
Started | 3 | 3 | 3 | 3 | 3 | 2 | 3 | 2 | 3 | 3 | 3 | 3
Completed | 3 | 3 | 3 | 3 | 3 | 2 | 3 | 2 | 3 | 3 | 3 | 3
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety analysis set: All subjects who received at least 1 dose of trial medication and who had follow-up safety assessments. As per Statistical Analysis Plan, Baseline Characteristics were to be reported for the overall population only. A summary by sequence or by some other grouping variable was not foreseen and thus is not available.
Groups:
- All Subjects: Subjects randomized to receive a single oral dose of MSC2499550A formulation at 20 milligram per kilogram (mg/kg) dispersed in water, current praziquantel (PZQ) formulation (Cysticide®) at 40 mg/kg with water under fed conditions; MSC2499550A formulation at 10 mg/kg or 30 mg/kg dispersed in water under fed condition; MSC2499550A formulation at 20 mg/kg dispersed in water under fasted condition; MSC2499550A formulation at 20 mg/kg directly disintegrated in the mouth without water under fed condition in one of the intervention periods.
Arm/Group | All Subjects
Number analyzed (Participants) | 36
Age, Continuous [Mean (Standard Deviation); unit: Years] | 26.3 (6.99)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 36

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Plasma Concentration-time Curve (AUC) From Time Zero to Infinity (AUC0-inf) Adj of L-Praziquantel (L-PZQ) After Dose Adjustment
Description: The AUC(0-inf) was estimated by determining the total area under the curve of the concentration versus time curve extrapolated to infinity.
Time Frame: Pre-dose, 0.5, 1.0, 1.5, 2.0, 2.5, 3.0, 3.5, 4.0, 4.5, 5.0, 5.5, 6.0, 8.0, 12.0, 16 and 24 hours post-dose
Population: PK population: all randomized subjects treated according to protocol without relevant violations with respect to factors likely to affect comparability of PK results & availability of AUC0-inf for MSC2499550A in periods 1 & 2. Number of "participants analyzed" below (Measured Values) reflects number of participants with non-missing values.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour*nanogram per milliliter (h*ng/mL)
Groups:
- Treatment A: Subjects received a single oral dose of MSC2499550A formulation at 20 milligram per kilogram (mg/kg) dispersed in water under fed condition in one of the intervention periods. There was a wash-out period of at least 7 days between each intervention period.
- Treatment B: Subjects received a single oral dose of current PZQ formulation (Cysticide®) at 40 mg/kg with water, under fed condition in one of the intervention periods. There was a wash-out period of at least 7 days between each of the intervention period.
- Treatment C1: Subjects received a single oral dose of MSC2499550A formulation at 10 mg/kg dispersed in water under fed condition in one of the intervention periods. There was a wash-out period of at least 7 days between each of the intervention period.
- Treatment C2: Subjects received a single oral dose of MSC2499550A formulation at 30 mg/kg dispersed in water under fed condition in one of the intervention periods. There was a wash-out period of at least 7 days between each of the intervention period.
- Treatment D: Subjects received a single oral dose of MSC2499550A formulation at 20 mg/kg dispersed in water in fasted condition in one of the intervention periods. There was a wash-out period of at least 7 days between each of the intervention period.
- Treatment E: Subjects received a single oral dose of MSC2499550A formulation at 20 mg/kg directly disintegrated in the mouth without water under fed conditions in one of the intervention periods. There was a wash-out period of at least 7 days between each of the intervention period.
Arm/Group | Treatment A | Treatment B | Treatment C1 | Treatment C2 | Treatment D | Treatment E
Number analyzed (Participants) | 36 | 36 | 17 | 17 | 35 | 36
hour*nanogram per milliliter (h*ng/mL) | 825.2 (101.0) | 2066.0 (64.7) | 216.7 (102.8) | 2324.9 (76.4) | 506.2 (100.0) | 954.5 (96.4)
Statistical Analysis 1: Comparison: Treatment A vs Treatment B; Test type: Superiority or Other; Ratio (%) = 39.9, 90% CI 2-sided [34.7 to 46.0] — Percentage of Geometric Least Squares (LS) Mean Ratio (Treatment A/Treatment B) is reported
Statistical Analysis 2: Comparison: Treatment A vs Treatment C1; Test type: Superiority or Other; Ratio (%) = 27.3, 90% CI 2-sided [22.5 to 33.2] — Percentage of Geometric LS Mean Ratio (Treatment C1/Treatment A) is reported
Statistical Analysis 3: Comparison: Treatment A vs Treatment C2; Test type: Superiority or Other; Ratio (%) = 260.2, 90% CI 2-sided [214.0 to 316.4] — Percentage of Geometric LS Mean Ratio (Treatment C2/Treatment A) is reported
Statistical Analysis 4: Comparison: Treatment A vs Treatment D; Test type: Superiority or Other; Ratio (%) = 167.1, 90% CI 2-sided [143.9 to 194.0] — Percentage of Geometric LS Mean Ratio (Treatment A/Treatment D) is reported
Statistical Analysis 5: Comparison: Treatment A vs Treatment E; Test type: Superiority or Other; Ratio (%) = 115.7, 90% CI 2-sided [99.8 to 134.1] — Percentage of Geometric LS Mean Ratio (Treatment E/Treatment A) is reported

2. Secondary Outcome: Time to Reach the Maximum Plasma Concentration (Tmax) of L-Praziquantel (L-PZQ)
Time Frame: Pre-dose, 0.5, 1.0, 1.5, 2.0, 2.5, 3.0, 3.5, 4.0, 4.5, 5.0, 5.5, 6.0, 8.0, 12.0, 16 and 24 hours post-dose
Population: The pharmacokinetic (PK) population included all randomized subjects who were treated according to the protocol without relevant protocol violations with respect to factors likely to affect the comparability of PK results and the availability of the primary target variable AUC0-inf for MSC2499550A in periods 1 and 2.
Measure: Median (Full Range); unit: hour
Arm/Group | Treatment A | Treatment B | Treatment C1 | Treatment C2 | Treatment D | Treatment E
Number analyzed (Participants) | 36 | 36 | 18 | 17 | 35 | 36
hour | 2.500 [0.50 to 4.50] | 2.500 [1.00 to 4.50] | 2.250 [1.00 to 4.50] | 3.000 [1.00 to 4.50] | 2.000 [0.50 to 4.50] | 4.000 [0.50 to 5.00]

3. Secondary Outcome: Time Prior to the First Measurable (Non-zero) Concentration (Tlag) of L-Praziquantel (L-PZQ)
Description: Time prior to the first measurable (non-zero) concentration (tlag) of drug L-PZQ
Time Frame: Pre-dose, 0.5, 1.0, 1.5, 2.0, 2.5, 3.0, 3.5, 4.0, 4.5, 5.0, 5.5, 6.0, 8.0, 12.0, 16 and 24 hours post-dose
Population: as for outcome 2
Measure: Median (Full Range); unit: hour
Arm/Group | Treatment A | Treatment B | Treatment C1 | Treatment C2 | Treatment D | Treatment E
Number analyzed (Participants) | 36 | 36 | 18 | 17 | 35 | 36
hour | 0.0 [0.0 to 0.0] | 0.0 [0.0 to 1.0] | 0.0 [0.0 to 0.0] | 0.0 [0.0 to 0.0] | 0.0 [0.0 to 0.0] | 0.0 [0.0 to 0.0]

4. Secondary Outcome: Area Under the Plasma Concentration-time Curve (AUC) From Time Zero to the Last Sampling Time at Which the Concentration is at or Above the Lower Limit of Quantification (AUC0-t) of L-Praziquantel (L-PZQ) After Dose Adjustment
Description: The AUC (0-t) was defined as the area under the plasma concentration versus time curve from time zero to time of last quantifiable concentration at or above the lower limit of quantification (AUC0-t) of L-PZQ.
Time Frame: Pre-dose, 0.5, 1.0, 1.5, 2.0, 2.5, 3.0, 3.5, 4.0, 4.5, 5.0, 5.5, 6.0, 8.0, 12.0, 16 and 24 hours post-dose
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour*nanogram per milliliter (h*ng/mL)
Arm/Group | Treatment A | Treatment B | Treatment C1 | Treatment C2 | Treatment D | Treatment E
Number analyzed (Participants) | 36 | 36 | 18 | 17 | 35 | 36
hour*nanogram per milliliter (h*ng/mL) | 791.0 (103.6) | 2010.7 (66.1) | 186.2 (107.5) | 2273.5 (77.9) | 464.7 (102.9) | 918.0 (98.7)

5. Secondary Outcome: Extrapolated Area Under the Concentration Time Curve (AUC) From Time Tlast to Infinity Given as Percentage From AUC0-inf (AUCextra) of L-Praziquantel (L-PZQ)
Description: Extrapolated AUC from time tlast to infinity given as percentage from AUC0-inf. AUCextra =(last predicted concentration [Clast pred] divided by terminal elimination rate constant [lambda z]) divided by AUC0-inf., where Clast pred is the last predicted concentration.
Time Frame: Pre-dose, 0.5, 1.0, 1.5, 2.0, 2.5, 3.0, 3.5, 4.0, 4.5, 5.0, 5.5, 6.0, 8.0, 12.0, 16 and 24 hours post-dose
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Percent extrapolated
Arm/Group | Treatment A | Treatment B | Treatment C1 | Treatment C2 | Treatment D | Treatment E
Number analyzed (Participants) | 36 | 36 | 17 | 17 | 35 | 36
Percent extrapolated | 3.40 (73.8) | 2.20 (65.2) | 6.62 (85.3) | 1.80 (72.7) | 5.81 (82.5) | 3.15 (66.5)

6. Secondary Outcome: Maximum Observed Concentration in Plasma (Cmax) of L-Praziquantel (L-PZQ) After Dose Adjustment
Time Frame: Pre-dose, 0.5, 1.0, 1.5, 2.0, 2.5, 3.0, 3.5, 4.0, 4.5, 5.0, 5.5, 6.0, 8.0, 12.0, 16 and 24 hours post-dose
Population: The PK population included all randomized subjects who were treated according to the protocol without relevant protocol violations with respect to factors likely to affect the comparability of PK results and the availability of the primary target variable AUC0-inf for MSC2499550A in periods 1 and 2.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter (ng/mL)
Arm/Group | Treatment A | Treatment B | Treatment C1 | Treatment C2 | Treatment D | Treatment E
Number analyzed (Participants) | 36 | 36 | 18 | 17 | 35 | 36
nanogram per milliliter (ng/mL) | 378.83 (114.1) | 727.27 (63.3) | 89.93 (92.2) | 1051.76 (83.6) | 131.06 (110.6) | 471.18 (99.5)

7. Secondary Outcome: Apparent Terminal Half-life (T1/2) of L-Praziquantel (L-PZQ)
Description: The apparent terminal half-life was calculated by dividing natural log 2 with lambda z (ln2/lambda Z); where lambda Z is the terminal rate constant.
Time Frame: Pre-dose, 0.5, 1.0, 1.5, 2.0, 2.5, 3.0, 3.5, 4.0, 4.5, 5.0, 5.5, 6.0, 8.0, 12.0, 16 and 24 hours post-dose
Population: as for outcome 1
Measure: Median (Full Range); unit: hour
Arm/Group | Treatment A | Treatment B | Treatment C1 | Treatment C2 | Treatment D | Treatment E
Number analyzed (Participants) | 36 | 36 | 17 | 17 | 35 | 36
hour | 2.984 [1.01 to 6.49] | 3.788 [1.44 to 10.1] | 1.059 [0.623 to 7.58] | 3.296 [1.82 to 5.46] | 2.801 [0.869 to 24.9] | 2.711 [0.452 to 6.65]

8. Secondary Outcome: Relative Bioavailability (Frel) of L-Praziquantel (L-PZQ)
Description: Relative bioavailability (Frel) was calculated for L-PZQ only (treatment A versus treatment B) using the formula: Frel = (AUC0-inf (test or Treatment A)/AUC0-inf (reference or treatment B)) multiplied by 100.
Time Frame: Pre-dose, 0.5, 1.0, 1.5, 2.0, 2.5, 3.0, 3.5, 4.0, 4.5, 5.0, 5.5, 6.0, 8.0, 12.0, 16 and 24 hours post-dose
Population: as for outcome 6
Measure: Geometric Mean (95% Confidence Interval); unit: Percentage bioavailability
Groups:
- Treatment A and B: Subjects received MSC2499550A formulation at 20 mg/kg dispersed in water as first or second intervention followed by current PZQ formulation (Cysticide®) at 40 mg/kg with water as second or first intervention under fed condition. There was a wash-out period of at least 7 days between each of the intervention period.
Arm/Group | Treatment A and B
Number analyzed (Participants) | 36
Percentage bioavailability | 40.075 [33.90 to 47.38]

9. Secondary Outcome: Apparent Terminal Elimination Rate Constant (Lambda Z) of L-Praziquantel (L-PZQ)
Description: The lambda z was calculated as the negative of the slope of the log-linear regression of the natural logarithm concentration-time curve during the terminal phase.
Time Frame: Pre-dose, 0.5, 1.0, 1.5, 2.0, 2.5, 3.0, 3.5, 4.0, 4.5, 5.0, 5.5, 6.0, 8.0, 12.0, 16 and 24 hours post-dose
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: per hour (1/hour)
Arm/Group | Treatment A | Treatment B | Treatment C1 | Treatment C2 | Treatment D | Treatment E
Number analyzed (Participants) | 36 | 36 | 17 | 17 | 35 | 36
per hour (1/hour) | 0.250 (53.9) | 0.181 (46.3) | 0.432 (88.6) | 0.206 (31.9) | 0.244 (62.3) | 0.264 (65.2)

10. Secondary Outcome: Apparent Total Body Clearance of Drug From Plasma (CL/f) of L-Praziquantel (L-PZQ)
Description: The CL/f of L-PZQ was a measure of the rate at which it was metabolized or eliminated by normal biological processes. Clearance obtained after oral dose was influenced by the fraction of the dose absorbed. The CL/F of L-PZQ from plasma was calculated using the formula: Dose divided by area under the concentration time curve from time zero to infinity (AUC0-inf).
Time Frame: Pre-dose, 0.5, 1.0, 1.5, 2.0, 2.5, 3.0, 3.5, 4.0, 4.5, 5.0, 5.5, 6.0, 8.0, 12.0, 16 and 24 hours post-dose
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter per hour
Arm/Group | Treatment A | Treatment B | Treatment C1 | Treatment C2 | Treatment D | Treatment E
Number analyzed (Participants) | 36 | 36 | 17 | 17 | 35 | 36
Liter per hour | 1665 (94.3) | 667.3 (60.1) | 3091 (92.9) | 923.5 (71.4) | 2729 (95.4) | 1440 (89.3)

11. Secondary Outcome: Apparent Volume of Distribution During the Terminal Phase (Vz/f) of L-Praziquantel (L-PZQ)
Description: The Vz/f was defined as the theoretical volume in which the total amount of L-PZQ required to uniformly distribute to produce the desired plasma concentration of L-PZQ. Apparent volume of distribution after oral dose (Vz/F) was influenced by the fraction absorbed. The Vz/f was calculated by dividing the dose with area under the concentration time curve from time zero to infinity multiplied with terminal elimination rate constant (lambda z) (Vz/f=Dose/( AUC0-inf* lambda z).
Time Frame: Pre-dose, 0.5, 1.0, 1.5, 2.0, 2.5, 3.0, 3.5, 4.0, 4.5, 5.0, 5.5, 6.0, 8.0, 12.0, 16 and 24 hours post-dose
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter
Arm/Group | Treatment A | Treatment B | Treatment C1 | Treatment C2 | Treatment D | Treatment E
Number analyzed (Participants) | 36 | 36 | 17 | 17 | 35 | 36
Liter | 6671 (62.9) | 3685 (62.8) | 7155 (72.4) | 4478 (62.8) | 11170 (81.1) | 5452 (62.4)

12. Secondary Outcome: Number of Subjects With Treatment Emergent Adverse Events (TEAEs) and Serious TEAEs, TEAEs Leading to Death and TEAEs Leading to Discontinuation
Description: An Adverse Event (AE) was defined as any new untoward medical occurrences/worsening of pre-existing medical condition without regard to possibility of causal relationship. A Serious Adverse Event (SAE) was an AE that resulted in any of the following outcomes: death; life threatening; persistent/significant disability/incapacity; initial or prolonged inpatient hospitalization; congenital anomaly/birth defect. TEAEs were adverse events that occurred between the first dose of study drug and up to 3-10 days after the last dose that were absent before treatment or that worsened relative to pretreatment state. Subjects who discontinued and who died due to TEAEs were also reported.
Time Frame: From the first dose of study drug administration up to 3-10 days after the last dose of the study drug (up to a maximum of 7 weeks)
Population: The safety analysis set consisted of all subjects who received at least one dose of the trial medication and who had follow-up safety assessments.
Measure: Number; unit: Subjects
Arm/Group | Treatment A | Treatment B | Treatment C1 | Treatment C2 | Treatment D | Treatment E
Number analyzed (Participants) | 36 | 36 | 18 | 17 | 35 | 36
Subjects
  TEAEs | 8 | 17 | 4 | 4 | 5 | 1
  Serious TEAEs | 0 | 0 | 0 | 0 | 0 | 0
  TEAEs leading to discontinuation | 0 | 0 | 0 | 0 | 0 | 0
  TEAEs leading to death | 0 | 0 | 0 | 0 | 0 | 0

13. Secondary Outcome: Palatability Score
Description: Each administration was assessed at 0 minutes on Day 1 for flavor, smell, sweetness, overall liking of the medicine and at 2-5 minutes on Day 1 for taste in mouth and acceptability to swallow using a modified 100 millimeter (mm), visual analog scale (VAS) incorporating a facial hedonic scale, where lower score (0) indicates "not acceptable/not liked at all" and higher score (100) indicates "very acceptable/liked very much".
Time Frame: 0 min for flavor, smell, sweetness, overall liking; 2-5 minutes post dose for taste in mouth and acceptability on Day 1
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: millimeter (mm)
Arm/Group | Treatment A | Treatment B | Treatment C1 | Treatment C2 | Treatment D | Treatment E
Number analyzed (Participants) | 36 | 36 | 18 | 17 | 35 | 36
millimeter (mm)
  Flavor: Day 1: 0 min | 67.5 (22.19) | 45.8 (24.04) | 72.2 (27.17) | 68.8 (22.33) | 65.9 (22.95) | 32.9 (29.10)
  Smell: Day 1: 0 min | 63.1 (21.63) | 56.4 (26.32) | 64.8 (25.22) | 61.9 (21.64) | 64.6 (19.67) | 46.9 (26.17)
  Sweetness: Day 1: 0 min | 74.8 (19.42) | 30.5 (20.80) | 72.2 (23.97) | 73.0 (19.31) | 68.0 (22.12) | 40.8 (30.59)
  Overall liking of Medicine: Day 1: 0 min | 67.8 (21.75) | 47.0 (28.22) | 69.7 (26.21) | 68.0 (20.47) | 63.3 (23.86) | 53.2 (26.10)
  Taste in Mouth: Day 1:2-5 minutes after medication | 50.9 (26.42) | 39.5 (26.12) | 68.9 (27.77) | 47.1 (28.29) | 47.7 (26.82) | 29.5 (26.12)
  Acceptable to swallow:Day1:2-5min after medication | 80.7 (17.57) | 59.2 (27.65) | 82.5 (23.04) | 68.7 (21.28) | 70.0 (19.50) | 38.1 (29.90)

14. Secondary Outcome: Number of Subjects With Clinical Significant Laboratory Abnormalities, Electrocardiogram (ECG), Physical Examination and Vital Signs Reported as Treatment Emergent Adverse Events
Description: Any clinically significant changes in laboratory evaluations ECGs,physical examination (body weight) and vital signs (temperature, blood pressure, pulse rate) were recorded as treatment emergent adverse events. Following parameters were analyzed for laboratory examination: hematology (haemoglobin, hematocrit, red blood cell count, mean cell hemoglobin [MCH], MCH concentration, mean cell volume, white cell count, platelets, neutrophils, lymphocytes, monocytes, eosinophils, Basophils); serum chemistry (sodium, potassium, calcium, inorganic phosphate, creatinine, total protein, albumin, urea, uric acid, aspartate aminotransferase [AST], alanine aminotransferase [ALT] gamma glutamyl transpeptidase, total bilirubin, alkaline phosphatase, glucose, triglycerides cholesterol); urinalysis (protein, glucose, ketones, pH, blood, leukocytes, nitrite); The 12-lead ECGs were recorded after the subjects had rested for at least 5 minutes in supine position.
Time Frame: as for outcome 12
Population: as for outcome 12
Measure: Number; unit: Subjects
Arm/Group | Treatment A | Treatment B | Treatment C1 | Treatment C2 | Treatment D | Treatment E
Number analyzed (Participants) | 36 | 36 | 18 | 17 | 35 | 36
Subjects
  Laboratory abnormalities | 0 | 0 | 0 | 0 | 0 | 0
  ECG abnormalities | 0 | 0 | 0 | 0 | 0 | 0
  Vital signs abnormalities | 0 | 0 | 0 | 0 | 0 | 0
  Physical signs abnormalities | 0 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Arm/Group | Treatment A | Treatment B | Treatment C1 | Treatment C2 | Treatment D | Treatment E
Serious Adverse Events (participants affected / at risk) | 0/36 | 0/36 | 0/18 | 0/17 | 0/35 | 0/36
Other Adverse Events (participants affected / at risk) | 8/36 | 17/36 | 4/18 | 4/17 | 5/35 | 1/36
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment A (N=36) | Treatment B (N=36) | Treatment C1 (N=18) | Treatment C2 (N=17) | Treatment D (N=35) | Treatment E (N=36)
Abdominal Discomfort (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0 | 0
Abdominal Pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Abdominal Pain Upper (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 1 | 1
Nausea (Gastrointestinal disorders) | 1 | 5 | 0 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 1 | 0 | 1 | 0 | 0 | 0
Influenza (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Tonsillitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Excoriation (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Dysgeusia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 6 | 11 | 0 | 2 | 5 | 0
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other